CLINICAL TRIAL: NCT02512978
Title: Thyroid Hormone Replacement for Hypothyroidism and Acute Myocardial Infarction
Brief Title: Thyroid Hormone Replacement for Hypothyroidism and Acute Myocardial Infarction(ThyroHeart-AMI)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); Peking Union Medical College Hospital (Other); Peking University Third Hospital (Other); Beijing Anzhen Hospital (Other); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); The Luhe Teaching Hospital of the Capital Medical University (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z15110700400000
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Myocardial Infarction; Hypothyroidism
Keywords: myocardial infarction; hypothyroidism; levothyroxine; cardiac magnetic resonance imaging; myocardial perfusion/metabolism radionuclide imaging; myocardial fibrosis; myocardial perfusion/metabolism; cardiac function
MeSH Terms: conditions — Myocardial Infarction; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levothyroxine group (Experimental): The patients allocated to levothyroxine group receive levothyroxine with a starting dose of 12.5ug.
  Interventions: Drug: Levothyroxine
- Standard therapy group (No Intervention): The patients in this group receive standard therapy in consistent with the local clinical practice.

INTERVENTIONS:
Drug: Levothyroxine — Levothyroxine is used to normalize the thyroid hormone level of patients allocated to levothyroxine.
  Other Names: Euthyrox
  Arms: Levothyroxine group

SUMMARY:
Based on accumulating evidences showing that hypothyroid status is associated with poor prognosis among acute myocardial infarction (AMI) patients, the study is designed to evaluate whether replacement treatment with levothyroxine could have beneficial effects on patients with AMI and hypothyroidism. This is a multicenter prospective computerized-randomized trial stratified by ejection fraction with a 1:1 ratio to levothyroxine group or standard therapy group.

DETAILED DESCRIPTION:
The primary hypothesis is that reversing the hypothyroid status with levothyroxine on top of standard therapy for AMI is safe and has beneficial effects on cardiac function, myocardial perfusion/metabolism and myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75, male or non-pregnant female;
2. Is diagnosed acute myocardial infarction and received primary percutaneous coronary intervention (PCI);
3. With presence of hypothyroid status (i.e., TSH >7.0 mIU/L and (or) fT3 <1.79 pg/mL);
4. Is able to understand the objective of the trial, takes part voluntarily and signs the written informed consent form.

Exclusion Criteria:

1. Those who have participated in other drug or therapeutic equipment clinical trials but do not reach the main study endpoint time limit;
2. Symptoms of severe heart failure (Killip Class III and above);
3. Severely impaired renal function before surgery: serum creatinine > 2.0mg/dl;
4. Impaired liver function before surgery: Serum GPT > 120U/L;
5. Those who have prior thyroid diseases and already on levothyroxine or anti-thyroid medicines;
6. Those taking medicine which can affect the test of thyroid function;
7. Patients who plan to undergo coronary artery bypass grafting or other surgery within 3 months;
8. Those having prior myocardial infarction;
9. Patients who are deemed by the researchers to have low compliance and unable to abide by the requirements and complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The improvement of Left Ventricular ejection fraction assessed by cardiac magnetic resonance imaging | within 6 months of patient enrolled

SECONDARY OUTCOMES:
Myocardial perfusion and metabolism detected by 99Tcm-MIBI SPECT and 18F-FDG PET imaging | Within 6 months of patient enrolled
  Patterns of myocardial perfusion/metabolism were classified as normal, mismatch, mild-moderate match and severe match
The severity of myocardial fibrosis assessed by late-gadolinium enhancement cardiac magnetic resonance imaging(cMRI-LGE) | Within 6 months of patient enrolled
Major adverse cardiac and cerebrovascular events | within 12 months of patient enrolled
  The composite endpoint of cardiac death, myocardial infarction, target vessel revascularization and cerebrovascular accident.
Death by any cause | Within 12 months of patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Cardiovascular Hospital, Beijing, China

REFERENCES:
- [Result] Li J, Li X, Wang Q, Hu S, Wang Y, Masoudi FA, Spertus JA, Krumholz HM, Jiang L; China PEACE Collaborative Group. ST-segment elevation myocardial infarction in China from 2001 to 2011 (the China PEACE-Retrospective Acute Myocardial Infarction Study): a retrospective analysis of hospital data. Lancet. 2015 Jan 31;385(9966):441-51. doi: 10.1016/S0140-6736(14)60921-1. Epub 2014 Jun 23. PMID 24969506
- [Result] Pingitore A, Chen Y, Gerdes AM, Iervasi G. Acute myocardial infarction and thyroid function: new pathophysiological and therapeutic perspectives. Ann Med. 2012 Dec;44(8):745-57. doi: 10.3109/07853890.2011.573501. Epub 2011 May 13. PMID 21568669
- [Result] Mourouzis I, Forini F, Pantos C, Iervasi G. Thyroid hormone and cardiac disease: from basic concepts to clinical application. J Thyroid Res. 2011;2011:958626. doi: 10.4061/2011/958626. Epub 2011 Jun 19. PMID 21765997
- [Result] Cakar M, Demirbas S, Demirkol S, Karaman M, Balta S, Unlu M. Chicken or egg? Which one is first? Myocardial infarction or low thyroid hormones? Intern Med. 2013;52(5):645. doi: 10.2169/internalmedicine.52.9285. Epub 2013 Mar 1. No abstract available. PMID 23448784
- [Result] Ceremuzynski L, Gorecki A, Czerwosz L, Chamiec T, Bartoszewicz Z, Herbaczynska-Cedro K. Low serum triiodothyronine in acute myocardial infarction indicates major heart injury. Kardiol Pol. 2004 May;60(5):468-80; discussion 473-4. English, Polish. PMID 15247962
- [Result] Chen YF, Kobayashi S, Chen J, Redetzke RA, Said S, Liang Q, Gerdes AM. Short term triiodo-L-thyronine treatment inhibits cardiac myocyte apoptosis in border area after myocardial infarction in rats. J Mol Cell Cardiol. 2008 Jan;44(1):180-7. doi: 10.1016/j.yjmcc.2007.09.009. Epub 2007 Oct 26. PMID 17964598
- [Result] Bai MF, Gao CY, Yang CK, Wang XP, Liu J, Qi DT, Zhang Y, Hao PY, Li MW. Effects of thyroid dysfunction on the severity of coronary artery lesions and its prognosis. J Cardiol. 2014 Dec;64(6):496-500. doi: 10.1016/j.jjcc.2014.03.009. Epub 2014 Jun 17. PMID 24951271
- [Result] Wang WY, Tang YD, Yang M, Cui C, Mu M, Qian J, Yang YJ. Free triiodothyronine level indicates the degree of myocardial injury in patients with acute ST-elevation myocardial infarction. Chin Med J (Engl). 2013 Oct;126(20):3926-9. PMID 24157158
- [Result] Zhang B, Peng W, Wang C, Li W, Xu Y. A low fT3 level as a prognostic marker in patients with acute myocardial infarctions. Intern Med. 2012;51(21):3009-15. doi: 10.2169/internalmedicine.51.7902. Epub 2012 Nov 1. PMID 23124142
- [Result] Mourouzis I, Giagourta I, Galanopoulos G, Mantzouratou P, Kostakou E, Kokkinos AD, Tentolouris N, Pantos C. Thyroid hormone improves the mechanical performance of the post-infarcted diabetic myocardium: a response associated with up-regulation of Akt/mTOR and AMPK activation. Metabolism. 2013 Oct;62(10):1387-93. doi: 10.1016/j.metabol.2013.05.008. Epub 2013 Jun 15. PMID 23773982
- [Result] Mourouzis I, Mantzouratou P, Galanopoulos G, Kostakou E, Roukounakis N, Kokkinos AD, Cokkinos DV, Pantos C. Dose-dependent effects of thyroid hormone on post-ischemic cardiac performance: potential involvement of Akt and ERK signalings. Mol Cell Biochem. 2012 Apr;363(1-2):235-43. doi: 10.1007/s11010-011-1175-9. Epub 2011 Dec 2. PMID 22134702
- [Result] Tang YD, Kuzman JA, Said S, Anderson BE, Wang X, Gerdes AM. Low thyroid function leads to cardiac atrophy with chamber dilatation, impaired myocardial blood flow, loss of arterioles, and severe systolic dysfunction. Circulation. 2005 Nov 15;112(20):3122-30. doi: 10.1161/CIRCULATIONAHA.105.572883. Epub 2005 Nov 7. PMID 16275864
- See also: heart attack — http://www.nlm.nih.gov/medlineplus/heartattack.html
- See also: hypothyroidism — http://www.nlm.nih.gov/medlineplus/hypothyroidism.html
- See also: levothyroxine — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a682461.html